CLINICAL TRIAL: NCT04301492
Title: Tolerability, Safety and Efficacy of Vortioxetine for Treatment od Depression in Parkinson's Disease: a 16 Week Open Label Study
Brief Title: Tolerability, Safety and Efficacy of Vortioxetine
Acronym: VorDe-PD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VorDe-PD; 2018-004112-21 (EudraCT Number)
Record Dates: First submitted 2020-02-17; First posted 2020-03-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Depression
Keywords: vortioxetine; tolerability; safety; parkinson's disease
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortioxetine (Experimental): first visit medical and pharmacological history will be collected and ECG, laboratory tests and clinical assessment will be performed. After verifying the absence of significant abnormalities at the ECG and laboratory tests and after confirming all inclusion and exclusion criteria, subjects will perform the second visit (Week 1 - Visit 2) to receive study drug (Brintellix drops 20 mg/ml). All subjects will be instructed to take Vortioxetine 1 drop every day after lunch, increasing of 1 drop per day arriving to 10 drops per day. After 5 days from the beginning of treatment, subject will be contacted by phone to check on tolerability and in absence of side effects, the dosage will be increased to 10 drops per day (Visit 3- Phone contact). At Week 4-8-12 (Visits 4-5-6) patients will return to the site to perform all clinical evaluations required and to receive study drug. Visit 7 subjects will return to the site to perform all the assessment required by protocol.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — 16 weeks for each participant. During the first visit a collection of medical and pharmacological history will be collected and ECG, laboratory tests and clinical assessment will be performed. After verifying the absence of significant abnormalities at the ECG and laboratory tests and after confirming all inclusion and exclusion criteria, subjects will perform the second visit to receive study drug (Brintellix drops 20 mg/ml). All subjects will be instructed to take Vortioxetine 1 drop every day after lunch, increasing of 1 drop per day arriving to 10 drops per day. After 5 days from the beginning of treatment, subject will be contacted by phone to check on tolerability and in absence of side effects, the dosage will be increased to 10 drops per day. At Week 4-8-12 patients will return to the site to perform all clinical evaluations required and to receive study drug.

SUMMARY:
Depression is a psychiatric disorder frequently found in Parkinson's disease (MP), affecting approximately 40-50% of patients and assuming the characteristics of major depression in 17% of cases. Vortioxetine is a new antidepressant, which inaugurates the class of "multimodal" antidepressants, able to exert modulation of serotonergic receptors, inhibit serotonin reuptake, modulate other neurotransmitters such as norepinephrine, dopamine, acetylcholine and histamine.

The primary endpoint of this study will be to verify safety and tolerability of vortioxetine in the treatment of sustained depression in PD. Safety will be assessed through the recording of treatment emergent adverse events (TEAE) and vital signs in each study visits and laboratory tests, ECG, physical and neurological examination at baseline and End of study. The non worsening of motor disability evaluated through Unified Parkinson's Disease Rating Scale (UPDRS) will be the tolerability end point.

The secondary endpoint will be to demonstrate the efficacy on depression: efficacy measures will include Hamilton Depression Rating Scale (HAM-D-17), Beck Depression Inventory (BDI), CGI-S and CGI-I.

DETAILED DESCRIPTION:
Depression is a psychiatric disorder frequently found in Parkinson's disease (MP), affecting approximately 40-50% of patients and assuming the characteristics of major depression in 17% of cases. Depression can also precede the onset of motor symptoms, playing an important role in the clinical course of the disease. Indeed, the presence of depression has been associated with greater disability, a more rapid cognitive decline, a higher mortality and a heavier burden for families and caregivers.The mechanisms underlying depression in MP are still not completely clarified, but autopsy and functional anatomy studies have demonstrated the presence of alterations in the limbic system and in noradrenergic and serotonergic nuclei of the brainstem.This dual nature accounts for the partial ineffectiveness of the common antidepressants that do not target alterations of the dopaminergic system.

Vortioxetine is a new antidepressant, which inaugurates the class of "multimodal" antidepressants, able to exert modulation of serotonergic receptors, inhibit serotonin reuptake, modulate other neurotransmitters such as norepinephrine, dopamine, acetylcholine and histamine.

Currently, tricyclic antidepressants and selective serotonin reuptake inhibitors represent the most common pharmacotherapy for depression treatment in PD patients. Although, they can induce or increase motor disability and other PD symptoms. It is of paramount importance finding a novel therapeutic approach able to positively impact on depression without worsening motor dysfunction. Therefore Vortioxetine can represent an innovative drug in the treatment of depression in PD thanks to its ability to increase dopaminergic neurotransmission in brain structures usually associated with depression.

This is a pilot, single centre, open label, ITT study which will be conducted at the l'IRCCS San Raffaele Pisana, under the responsibility of Fabrizio Stocchi, Principal Investigator.

The study will be conducted in accordance with the guidelines for Good Clinical Practice, in line with the law on the processing of patients' personal data and the principles of the Helsinki Declaration.

Patients will receive informed consent before they are included in the study.

Study population will include patients with idiopathic Parkinson's disease in stage I-III of the disease, suffering from sustained depression. 20 consecutive PD outpatient referred to the center for the study of Parkinson's disease and movement disorders of the IRCCS San Raffaele Pisana will be enrolled.

Since this is a pilot, monocentric study, calculation of the sample size is not required.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female of every ethnic group, age 30 to 80 years

  * Diagnosis of Parkinson's disease according UK Brain Bank Criteria
  * Hoehn &Yahr: stage 1 to 3
  * Patients with diagnosis of sustained depression
  * Hamilton Depression Rating Scale score (HAM-D-17) ≥ 14
  * Beck Depression Inventory score (BDI)≥13
  * Stable doses of antiparkinsonian drugs for at least 4 weeks.
  * Patients able to understand and provide written informed consent
  * Female patients in post-menopausal state with at least one year absence of vaginal bleeding or spotting or be surgically sterile
  * Women of childbearing potential must use an acceptable method of contraception
  * Men with a potentially fertile partner must have had a vasectomy or be willing to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* • Atypical Parkinsonism.

  * Subjects at risk of suicide (with a score ≥ 3 at the Item 3 of the HAM-D-17)
  * Any significant psychiatric, metabolic and systemic significant concomitant disease
  * Patients with clinically significant out of range laboratory values
  * Patients with history of epileptic seizures
  * Subjects with Dopa Dysregulation Syndrome (DDS)
  * Subjects treated with irreversible IMAO and IMAO-A
  * Use of vortioxetine in the past 30 days
  * Patient treated with oral anticoagulant
  * Patients participating in a clinical trial in the last 6 weeks
  * Patients with moderate-severe cognitive decline not able to provide consent form
  * Patients currently lactating or pregnant or planning to become pregnant during the duration of the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  The primary endpoint of this study will be to verify tolerability and safety of vortioxetine in the treatment of sustained depression in PD. The non worsening of motor disability evaluated through Unified Parkinson's Disease Rating Scale (UPDRS) will be the tolerability end point.

SECONDARY OUTCOMES:
Incidence of Vortioxetine in the decrease of depression | through study completion, an average of 1 year
  The secondary endpoint will be to demonstrate the efficacy on depression: efficacy measure will include Hamilton Depression Rating Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS San Raffaele, Roma
  - IRCCS San Raffaele Roma, Rome

IPD SHARING:
Plan to Share IPD: Yes
after the end of sudy
Supporting Information: Study Protocol
Time Frame: after the end of study
Access Criteria: request by email